CLINICAL TRIAL: NCT00273299
Title: A 6-Week Study to Evaluate the Combination of Valsartan/HCTZ (160/12.5mg With Forced Titration to Maximum Dose of 320/25mg) Compared to Valsartan Monotherapy (160mg With Forced Titration to 320mg) as Initial Therapy in Patients With Severe Hypertension
Brief Title: Valsartan/Hydrochlorothiazide Combination in the Treatment of Severe Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAH631D2301
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Hypertension
Keywords: hypertension; high blood pressure; valsartan/hydrochlorozide; severe hypertension
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Hydrochlorothiazide

INTERVENTIONS:
Drug: valsartan plus hydrochlorothiazide

SUMMARY:
The purpose of this study is to assess the potential of using valsartan/HCTZ as initial therapy in patients with severe hypertension compared to valsartan alone as initial therapy, and to determine whether a greater proportion of patients achieve blood pressure control with the combination compared to the monotherapy without producing an unacceptable adverse event profile.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed severe hypertension

Exclusion Criteria:

* Inability to discontinue all prior antihypertensive medications
* Heart failure of any kind
* History of stroke, transient ischemic attack, myocardial infarction, chest pain, abnormal heart rhythm Liver, kidney, or pancreas disease
* Diabetes with poor glucose control
* Allergy to certain medications used to treat high blood pressure

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2005-11; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Blood pressure less than 140/90 mmHg after 4 weeks

SECONDARY OUTCOMES:
Blood pressure less than 140/90 mmHg after 6 weeks
Diastolic blood pressure less than 90 mmHg after 4 and 6 weeks
Systolic blood pressure less than 140 mmHg after 4 and 6 weeks
Change from baseline in systolic and diastolic blood pressure after 4 and 6 weeks
Adverse events and serious adverse events at each study visit for 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Calhoun DA, Glazer RD, Pettyjohn FS, Coenen PD, Zhao Y, Grosso A. Efficacy and tolerability of combination therapy with valsartan/hydrochlorothiazide in the initial treatment of severe hypertension. Curr Med Res Opin. 2008 Aug;24(8):2303-11. doi: 10.1185/03007990802271946. Epub 2008 Jun 28. PMID 18593517